CLINICAL TRIAL: NCT03243825
Title: Comparative Study of Neoadjuvant Chemo/Brachytherapy and Chemotherapy Alone Before Radical Hysterectomy in Stage Ib2-IIa2 Cervical Cancer
Brief Title: Comparative Study of Different Neoadjuvant Therapies Before Radical Hysterectomy in Stage Ib2-IIa2 Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ning Li, Doctor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2012B38
Record Dates: First submitted 2014-07-27; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cervical Cancer
Keywords: neoadjuvant chemotherapy; brachytherapy; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemo/brachytherapy (Experimental): Patients in this arm will receive neoadjuvant chemotherapy (paclitaxel/cisplatinum) and brachytherapy before radical hysterectomy.
  Interventions: Radiation: combination group
- chemotherapy (Active Comparator): Patients in this arm will receive neoadjuvant chemotherapy (paclitaxel/cisplatinum) before radical hysterectomy.
  Interventions: Drug: chemotherapy group

INTERVENTIONS:
Radiation: combination group — chemotherapy (paclitaxel/cisplatinum) and brachytherapy
  Arms: chemo/brachytherapy
Drug: chemotherapy group — chemotherapy: (paclitaxel/cisplatinum)
  Arms: chemotherapy

SUMMARY:
For stage Ib2-IIa2 cervical cancer patients, neoadjuvant therapy followed by radical hysterectomy and pelvic lymphadenectomy is one of the managements. Post-operative concurrent chemo-radiotherapy is necessary if the patients have high-risk factors, including positive surgical margin, parametrium and pelvic nodes. Our previous retrospective study showed that combination of neoadjuvant chemotherapy and brachytherapy reduced the proportion of post-operative concurrent chemo-radiotherapy compared to neoadjuvant chemotherapy alone.

DETAILED DESCRIPTION:
In the present study, the patients with stage Ib2-IIa2 cervical cancer will receive either neoadjuvant chemo/brachytherapy or neoadjuvant chemotherapy before radical hysterectomy and pelvic+/- para-aortic lymph node dissection. According to the surgical findings, post-operative chemo-radiotherapy will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed cervical cancer
* Clinical stage Ib2 or IIa2 (FIGO 2009)

Exclusion Criteria:

* Patients who not suitable for surgery
* Personal history of pelvic radiotherapy

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
proportion of post-operative chemo-radiotherapy | 2 months

SECONDARY OUTCOMES:
3-year disease-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Acadamy of Medical Sceinces, Beijing, China